CLINICAL TRIAL: NCT04200222
Title: Analyses of Maternal Plasma Cadmium, Lead and Vanadium Levels in the Diagnosis and Severity of Late-onset Preeclampsia; A Prospective and Comparative Study From Turkey
Brief Title: Vanadium in Late-onset Preeclampsia
Acronym: Vanadium PE
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH1
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preeclampsia: The diagnosis of L-PrE, as defined by the Committee on Terminology of the American College of Obstetricians and Gynecologists (ACOG), is established based on the presence of proteinuria (urinary excretion of protein ≥300 mg in a 24-h urine specimen, or proteinüria ≥1+ in dipstick) and a blood pressure level of ≥90/140 mmHg (two blood pressure measurements 6 h apart) that occurs after 34 weeks of gestation in a previously normotensive woman. The diastolic and/or systolic blood pressure <110/160 mm Hg, it was accepted as mild; and in case these values exceeded this level, it was accepted as severe. The study population consisted of 50 late-onset preeclampsia patients as study group and 50 patients with normal pregnancies as control group.
  Interventions: Diagnostic Test: cadmium, lead and vanadium measurements and compare
- Control: Pregnant women with uncomplicated pregnancies were randomly selected to serve as controls. Healthy subjects who had a normal pregnancy and outcomes without any fetal-neonatal complications were accepted into the control group.
  Interventions: Diagnostic Test: cadmium, lead and vanadium measurements and compare

INTERVENTIONS:
Diagnostic Test: cadmium, lead and vanadium measurements and compare — The method developed by Aliyev et al. was used for preparing the samples for analysis (1).
  The three metals (cadmium, lead and vanadium) were measured using inductively coupled plasma-mass spectrometry (Thermo Scientific ICAPQc, USA).
  1. Ovayolu A, Ovayolu G, Karaman E, Yuce T, Ozek MA, Turksoy VA. Amniotic fluid levels of selected trace elements and heavy metals in pregnancies complicated with neural tube defects. Congenit Anom (Kyoto). 2019:10.1111/cga.12363.

SUMMARY:
Introduction: Cadmium, lead and vanadium important pollutants produced from anthropogenic activities, has been suggested to be embryotoxic and fetotoxic in a lot of studies. However, the causes of preeclampsia are little known and heavy metals merit further investigation. We tested whether late-onset preeclampsia (L-PrE) was associated with exposure to these metals.

Methods: This study was designed to determine maternal plasma cadmium, lead and vanadium concentrations in women with L-PrE (n=46) compared to those of normotensive women (n=46). These three heavy metals concentrations measured using inductively coupled plasma-mass spectrometry were compared.

DETAILED DESCRIPTION:
This observational case-control study was conducted at the Department of Obstetrics and Gynecology, Cengiz Gokcek Public Hospital, Gaziantep, Turkey, between March 2018 and June 2019. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (reference no: 2019/36). The study strictly adhered to the principles of the Declaration of Helsinki. All subjects included in the study gave oral and written informed consent. Ninety-two women were enrolled in the study in two groups.

Data collection and Study intervention:

The diagnosis of L-PrE, as defined by the Committee on Terminology of the American College of Obstetricians and Gynecologists (ACOG), is established based on the presence of proteinuria (urinary excretion of protein ≥300 mg in a 24-h urine specimen, or proteinüria ≥1+ in dipstick) and a blood pressure level of ≥90/140 mmHg (two blood pressure measurements 6 h apart) that occurs after 34 weeks of gestation in a previously normotensive woman. The diastolic and/or systolic blood pressure <110/160 mm Hg, it was accepted as mild; and in case these values exceeded this level, it was accepted as severe. Every women in the study population underwent obstetric ultrasound examination and fetal-maternal assesment was carried out by one of the authors. The obstetric anamnesis were obtained from all subjects. The dempograhic data like age, gravidity, parity, body mass index (BMI) and gestational age were recorded. The gestational age was determined by calculation from the last menstrual period and supported by the ultrasonography measurements at first trimester of gestation. Maternal venous plasma samples were taken for measurement of cadmium, lead and vanadium levels after the diagnosis of L-PrE in outpatient clinic. These samples quickly centrifuged at 1,500 g for 10 min, plasma samples were seperated and stored at -80 C until the day of measurement. All patients with L-PrE were also hospitalized and their pregnancies were terminated. The samples of the control groups were obtained during the routine obstetrical care examination in the third trimester of pregnancy. Then, these pregnant women were followed-up until the delivery. Both groups were compared in terms of maternal age, BMI, week of gestation, gravida, parity, live born, systolic/diastolic blood pressure, total protein in spot urine sample, hemoglobin, hematocrit, platelet count, white blood cell count, urea, uric acid, albümin, blood urea nitrogen, creatinine, liver function tests (AST, ALT), lactic acid dehydrogenase, cadmium, lead and vanadium concentrions and infant weight at delivery. Small for gestational age (SGA) neonate was defined as birth weight <10th percentile for gestational age with Turkey's national nomogram as the reference for fetal growth. The samples were transferred within boxes in ice molds to Yozgat Bozok University Science and Technology Application and Research Center (Occupational and Environmental Toxicology Laboratory) for measuring heavy metal and trace element levels. The frequency of seafood consumption was divided into four categories: 2-3 per week, 1-2 per week, 1-2 per month, and rare. Smoking was classified into 3 groups (none, formerly smoker, and active smoking). Passive smoking was also categorized into 2 groups (no and yes). The education levels was classified into 4 groups (illiterate, primary education, high school, and university). The residences of women was classified as rural and urban. Furthermore, the residences of women have divided either living near a busy street (around 100 metres) or not.Small for gestational age (SGA) neonate was defined as birth weight <10th percentile for gestational age with Turkey's national nomogram as the reference for fetal growth.

The method developed by Aliyev et al. was used for preparing the samples for analysis One milliliter of plasma samples was placed into high-temperature-resistant Teflon tubes in a microwave oven, and 5 mL Suprapur® (Merck, Darmstadt, Germany) nitric acid (HNO3) and 5 mL ultra-pure water was added. All plasma samples were digested using a microwave digestion system (Start D; Milestone, MD, USA). After digestion, each sample was made to a total volume of 20 mL with 9 mL ultra-pure water in a 50 mL polypropylene tube. Nitric acid (Suprapur®, 65%) was used for digestion of samples and standard reference material. Ultra-pure water (Direct-Q®; Millipore, Darmstadt, Germany) was used for dilution of the standard (multi-element standard Chem-Lab, Zedelgem, Belgium) and sample preparations.

The three metals (cadmium, lead and vanadium) were measured using inductively coupled plasma-mass spectrometry (Thermo Scientific ICAPQc, USA). The operating parameters were set as follows: radiofrequency power 1550 W, nebulizer gas 0.96 L/min, plasma gas 0.88 L/min, nebulizer pressure 3.01 bar, dwell time 0.01 milliseconds, and spray chamber temperature 3.7°C. The sampler probe was washed between injections by rinsing with ultrapure water for 30 s, followed by washing with 2% HNO3 for 45 s, and finally rinsing with ultrapure water for 45 s. After the washing steps, the instrument automatically ran the next sample. An 11-point calibration curve (0.5-500 µg/L) was used to measure the level of each element. The r2 values of the calibration curves of all metals were calculated, and the minimum value was 0.9994. To ensure the accuracy of the results, each measurement of the samples and standards was repeated three times. The results of these measurements showed that the relative standard deviation (RSD) did not exceed 5%. Certified Reference Material (CRM-Seronorm™ Trace Elements Whole Blood L-2, Sero AS, Billingstad, Norway) was used for the validation method. To check the stability and sensitivity of the instrument, a mixture of internal standards (Hf) was used, and the mean and RSD values of metals were also calculated. The variations of each measurement of the quality controls was <15%. The relative percentage differences in replicate analyses were <5% in the samples and standards.

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia
* healthy pregnancy

Exclusion Criteria:

1. pregnant women with any systemic condition (such as chronic hypertension, renal disease and )
2. using any kind of medication/supplement intake throughout pregnancy (such as heparin)
3. history of medication for PE treatment at the time of first admission
4. smoking
5. drug user
6. patients who had fetal congenital abnormalities or genetic syndromes
7. multiple-gestation pregnancies
8. pregnancies resulting from in vitro fertilization
9. intrauterine fetal death
10. having family history of preeclampsia

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Preeclampsia, is a pregnancy complication characterized by high blood pressure and signs of damage to another organ system, most often the liver and kidneys. Preeclampsia usually begins after 20 weeks of pregnancy in women whose blood pressure had been normal. Late-onset preeclampsia is usually defined as preeclampsia that develops after 34 weeks of gestation.
Study Population: The investigators consecutively recruited 50 subjects with preeclampsia, and 50 healthy pregnancies selected for the control group.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome in these analyses was to compare cadmium, lead and vanadium levels in L-PrE group and control group. | 3 months
  The primary outcome in these analyses was to compare cadmium, lead and vanadium levels in L-PrE group and control group.

SECONDARY OUTCOMES:
The secondary outcome was to compare the cadmium, lead and vanadium levels in mild L-PrE group and severity L-PrE group. | 1 day
  The secondary outcome was to compare the cadmium, lead and vanadium levels in mild L-PrE group and severity L-PrE group.

OTHER OUTCOMES:
Tertiary outcome was to compare the cadmium, lead and vanadium levels in SGA group and non-SGA group. | 1 day
  Tertiary outcome was to compare the cadmium, lead and vanadium levels in SGA group and non-SGA group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gruzewska K, Michno A, Pawelczyk T, Bielarczyk H. Essentiality and toxicity of vanadium supplements in health and pathology. J Physiol Pharmacol. 2014 Oct;65(5):603-11. PMID 25371519
- [Background] Wang F, Fan F, Wang L, Ye W, Zhang Q, Xie S. Maternal Cadmium Levels During Pregnancy and the Relationship with Preeclampsia and Fetal Biometric Parameters. Biol Trace Elem Res. 2018 Dec;186(2):322-329. doi: 10.1007/s12011-018-1312-3. Epub 2018 Apr 12. PMID 29651732
- [Background] Zhang Q, Huang Y, Zhang K, Huang Y, Yan Y, Wang F, Wu J, Wang X, Xu Z, Chen Y, Cheng X, Li Y, Jiao J, Ye D. Cadmium-induced immune abnormality is a key pathogenic event in human and rat models of preeclampsia. Environ Pollut. 2016 Nov;218:770-782. doi: 10.1016/j.envpol.2016.07.073. Epub 2016 Aug 7. PMID 27511439
- [Background] Ovayolu A, Ovayolu G, Karaman E, Yuce T, Ozek MA, Turksoy VA. Amniotic fluid levels of selected trace elements and heavy metals in pregnancies complicated with neural tube defects. Congenit Anom (Kyoto). 2020 Sep;60(5):136-141. doi: 10.1111/cga.12363. Epub 2019 Nov 27. PMID 31743503
- [Result] Poropat AE, Laidlaw MAS, Lanphear B, Ball A, Mielke HW. Blood lead and preeclampsia: A meta-analysis and review of implications. Environ Res. 2018 Jan;160:12-19. doi: 10.1016/j.envres.2017.09.014. Epub 2017 Sep 21. PMID 28938191

DOCUMENTS (1):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04200222/Prot_000.pdf